CLINICAL TRIAL: NCT07091968
Title: Pilot Feasibility Trial to Evaluate a Technology-Enabled Approach to Enhance Depression Referral Uptake Among Cancer Survivors
Brief Title: Feasibility of a Technology-Based Intervention for Depression Referral Uptake in Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Katherine Sterba, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00142801
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Depression
MeSH Terms: conditions — Neoplasms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-Enabled Tailored Referral (Experimental): Participants in the intervention arm will receive a technology-enabled, text-based referral platform designed to improve depression referral uptake. The platform includes an initial text with a brief video explaining common barriers, tailored text messages based on participant-identified barriers, and an automated referral link. Messages are mapped to stages of readiness using the Transtheoretical Model and sent every two days over a two-week period to non-responders or decliners. This approach aims to engage survivors with depression care through personalized, accessible, and stage-matched communication.
  Interventions: Behavioral: Technology-Enabled Tailored Referral
- Usual Care Referral (No Intervention): Participants in the usual care arm will receive a printed flyer with information on local and virtual mental health treatment resources. The flyer includes contact details for emergency services, psychiatric urgent care, psychological oncology programs, support groups, and behavioral health clinics in the Charleston area, many of which offer telehealth options. No personalized messages or follow-up outreach will be provided.

INTERVENTIONS:
Behavioral: Technology-Enabled Tailored Referral — Participants in the intervention arm will receive a technology-enabled, text-based referral platform designed to improve depression referral uptake. The platform includes an initial text with a brief video explaining common barriers, tailored text messages based on participant-identified barriers, and an automated referral link. Messages are mapped to stages of readiness using the Transtheoretical Model and sent every two days over a two-week period to non-responders or decliners. This approach aims to engage survivors with depression through personalized, accessible, and stage-matched communication.
  Arms: Technology-Enabled Tailored Referral

SUMMARY:
Depression is very common in cancer survivors but there are challenges to linking those in need of treatment efficiently to care. In this study, investigators will test the feasibility and acceptability of a new text-based approach to connect cancer survivors with depression with care.

DETAILED DESCRIPTION:
The objectives of this study are 1) to evaluate the feasibility and acceptability of a technology-enabled approach to improve referral uptake among cancer survivors and 2) to evaluate the preliminary efficacy of this approach to improve referral uptake compared to usual care among cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diagnosis of cancer
* upcoming appointment in an HCC or HCN oncology clinic within 14 days
* English proficiency
* ownership of a cellphone with SMS text capability.
* elevated depressive symptoms at screening (as measured by > 3 on the PHQ-2)

Exclusion Criteria:

* cognitive impairment as evaluated by attending physician
* currently receiving counseling for depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability | 6 weeks
  The co-primary outcomes are acceptability and feasibility of the technology-enabled referral intervention. Acceptability will be measured using the System Usability Scale (SUS) at 6 weeks, with a score ≥80 indicating high acceptability. Feasibility will be assessed by determining whether key components of the intervention were successfully delivered and engaged with over the course of the 4 week intervention, including: (1) initiation of text-based contact, (2) delivery of tailored messages, and (3) access of the automated referral link by the participant. Additionally, participant engagement will be evaluated by tracking whether they opened the initial message, viewed the embedded video, and read the tailored text messages. These outcomes will be summarized using a Bayesian beta-binomial approach to determine go/no-go decision thresholds for future scale-up.

SECONDARY OUTCOMES:
Referral Uptake | 6 weeks
  Referral uptake is defined as whether a participant initiates a mental health treatment referral at 6 weeks. It will be measured through participant self-report and, when available, verified via electronic health records or provider confirmation.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sterba, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Results will not be shared with individual participants; data will be used for internal analysis and publication.